CLINICAL TRIAL: NCT01147809
Title: A Randomized, Blinded, Placebo-controlled, Two-Phase, Sequential Cohort, Dose Finding Study to Assess the Safety and Efficacy of an Oral Thrombopoietin Receptor Agonist, Eltrombopag (SB-497115-GR), Administered to Patients With Solid Tumors Receiving Gemcitabine Monotherapy or the Combination of Gemcitabine Plus Carboplatin or Cisplatin
Brief Title: Safety and Efficacy Study for Solid Tumor Patients Treated With Eltrombopag
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 112765
Record Dates: First submitted 2010-05-20; First posted 2010-06-22 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Thrombocytopaenia
Keywords: Solid Tumor; Eltrombopag; chemotherapy-induced thrombocytopenia; Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eltrombopag (Active Comparator): Drug: eltrombopag olamine thrombopoietin receptor agonist
  Interventions: Drug: Eltrombopag olamine
- Placebo (Placebo Comparator): Other: Placebo Placebo tablets with no active pharmaceutical ingredient
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Eltrombopag olamine — thrombopoietin receptor agonist
  Arms: Eltrombopag
Other: Placebo — Placebo tablets with no active pharmaceutical ingredient
  Arms: Placebo

SUMMARY:
The present study is a randomized, blinded, placebo-controlled, two-Phase, sequential cohort, dose finding study to assess the safety and efficacy of eltrombopag in patients with solid tumors receiving gemcitabine monotherapy or the combination of gemcitabine plus carboplatin or cisplatin. Phase I of the study will examine safety and tolerability of various doses of eltrombopag to identify a dose and schedule of eltrombopag. Phase II will confirm that the chosen dose and schedule of eltrombopag from Phase I can deliver clinically meaningful benefit(s) to thrombocytopenic patients by improving platelet numbers.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria Subjects eligible for enrolment in Phase I and II of the study must meet all of the following criteria:

* Signed written informed consent.
* Age ≥ 18 years.
* Subjects with confirmed solid tumor and scheduled to receive at least two cycles of either gemcitabine monotherapy OR gemcitabine in combination with carboplatin or cisplatin at the same dosages and schedule in the study. Novel anticancer agents (e.g. bevacizumab, erlotinib) may be allowed if considered a standard treatment by the investigator. Subjects with only ONE current diagnosis of primary solid tumor will be allowed into the study.
* Note: For patients scheduled to receive any novel anticancer agents (e.g. bevacizumab, erlotinib), consultation and approval from the GSK medical monitor should occur before the subject is enrolled into the study.
* Life expectancy of at least 3 months, in the opinion of the investigator.
* ECOG-Zubrod performance status ≤ 2
* For Phase I: Pre-chemotherapy platelet count ≤ 300 Gi/L in the screening period before the subject start their first planned cycle of treatment with gemcitabine monotherapy OR gemcitabine in combination with carboplatin or cisplatin in the study.
* For Phase II (Part 1 and 2): Subjects must meet one of the following platelet count entry criteria:

  1. Subjects have not started the first cycle in this disease setting and have a platelet count < 150 Gi/L in the screening period as measured within 3 days before Day -5, OR
  2. Subjects started chemotherapy for this disease setting and had platelet count < 150 Gi/L on Day 1 in the preceding cycle before entry into the study, OR
  3. Platelet count < 100 Gi/L at Day 8 in the preceding cycle before entry into the study, OR
  4. Platelet count < 100 Gi/L at Day 15 in the preceding cycle before entry into the study (for subjects receiving Gemcitabine monotherapy) Note: For any of these platelet counts, a repeated platelet count may be allowed only once to ensure that the subject meets the above platelet count criteria and the latest count will be taken for the assessment of eligibility to the study..
* Subjects with previous chemotherapy treatment in a previous disease setting are allowed provided they have recovered from chemotherapy related toxicity except alopecia (and the lab parameters mentioned in Inclusion criteria in #9).
* Adequate organ function during screening period defined by the criteria below (adequate baseline organ function):
* SYSTEM LABORATORY VALUES
* Hematologic
* Platelets, see Inclusion criteria
* ANC (absolute neutrophil count) ≥1.5 × 109/L
* Hemoglobin ≥9 g/dL
* Prothrombin time (PT/INR) and activated partial thromboplastin time (aPTT) Within 80 to 120% of the normal range
* Hepatic
* Albumin ≥2.5 g/dL
* Serum bilirubin ≤1.5 x ULN AST and ALT

  * 3 × ULN without liver metastases
  * 5 × ULN if documented liver metastases
* Renal
* Serum Creatinine ≤ 1.2 x ULN
* Subjects with AST, ALT or bilirubin values outside the range(s) in the table due to Gilbert's syndrome or asymptomatic gall stones are not excluded.
* Women of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to randomization and agree to use effective contraception, during the study and for 4 weeks following the last dose of investigational product.
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from 2 weeks prior to randomization until 13 weeks after the last dose of study treatment.
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Lactating females.
* Pre-existing cardiovascular disease (congestive heart failure, New York Heart Association [NYHA] Grade III/IV), or arrhythmia known to increase the risk of thromboembolic events (e.g. atrial fibrillation), unstable angina, or subjects with a QTc >450 msec (QTc >480 msec for subjects with Bundle Branch Block) at study entry, or myocardial infarction within the preceding 6 months. Subjects with a34 pacemaker or defibrillator are not excluded provided that their cardiac function is within normal ranges.
* Note: For patients with pre-existing NYHA Grade II cardiovascular disease, the investigator should consult with GSK medical monitor before enrolling the subject into the study.
* Patients with known factor V leiden, antiphospholipid antibody syndrome, prothrombin gene mutations, ATIII deficiency, protein C deficiency, protein S deficiency OR recent history of arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism) within the preceding 6 months.
* Note: for patients with known risk factors for thromboembolism e.g., diabetes, hypercholesterolemia, recent major surgery etc., the investigator should consult with GSK medical monitor before enrolling the patient into the study and all risk factors should be documented in the CRF.
* Prior surgery within two weeks before study randomization or radiotherapy (RT) within four weeks before study randomization. Subjects with prior surgery or RT are not permitted into the study unless they have completely recovered from surgery and/or acute RT toxicity except for alopecia.
* Note: Note: patients with minor surgeries or outpatient procedures (e.g. insertion of central venous catheter) are immediately allowed in the study provided that there were no complications from the procedure or surgery.
* History of prior radiotherapy to more than 20% bone marrow bearing sites.
* History of platelet agglutination abnormality, platelet disorders or dysfunction or bleeding disorder that prevents reliable measurement of platelet counts.
* Subjects with a history of CNS metastases or clinical signs or symptoms of brain and/or leptomeningeal metastases confirmed by CT or MRI brain scan unless properly treated. Subjects with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to randomization will be excluded.
* Treated brain metastases are defined
* Having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed.
* Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician.

Note: if subject has performed a CT scan immediately prior to the screening period and CT could not be repeated, an MRI should be performed in the screening period to exclude the development of brain metastases and/or the progression of the pre-existing brain metastatic lesion(s).

* Administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of investigational product in the study. Concurrent participation in another interventional clinical trial or administration of any investigational drug during the study is also not permitted.
* A known immediate or delayed hypersensitivity reaction or idiosyncrasy that, in the opinion of the Investigator or GSK Medical Monitor is due to drugs chemically related to eltrombopag or excipients (e.g. mannitol).
* Subjects with known Hepatitis B, hepatitis C or Human Immunodeficiency Virus (HIV). Subjects with Gilbert's Syndrome are permitted into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-06; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (77):
- United States (32):
  - GSK Investigational Site, Sedona, Arizona
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Rancho Cucamonga, California
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Rome, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Bend, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Wynnewood, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Edmonds, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Vancouver, Washington
  - GSK Investigational Site, Yakima, Washington
- Belgium (4):
  - GSK Investigational Site, Charleroi
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Libramont
  - GSK Investigational Site, Namur
- Canada (2):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Toronto, Ontario
- Czechia (2):
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- Finland (2):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Tampere
- Germany (8):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Goslar, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Thessaloniki
- Hungary (5):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Kaposvár
  - GSK Investigational Site, Törökbálint
  - GSK Investigational Site, Zalaegerszeg
- India (2):
  - GSK Investigational Site, Madurai
  - GSK Investigational Site, Pune
- Ireland (2):
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Tallaght, Dublin
- Israel (6):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Tel Aviv
  - GSK Investigational Site, Zrifin
- Italy (5):
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Aviano (PN), Friuli Venezia Giulia
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Pisa, Tuscany
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Konin
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan

REFERENCES:
- [Derived] Winer ES, Safran H, Karaszewska B, Richards DA, Hartner L, Forget F, Ramlau R, Kumar K, Mayer B, Johnson BM, Messam CA, Mostafa Kamel Y. Eltrombopag with gemcitabine-based chemotherapy in patients with advanced solid tumors: a randomized phase I study. Cancer Med. 2015 Jan;4(1):16-26. doi: 10.1002/cam4.326. Epub 2014 Aug 28. PMID 25165041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) with solid tumors receiving gemcitabine monotherapy or the combination of gemcitabine plus carboplatin or cisplatin were eligible for enrollment into the study. The study comprised of 2 phases (I & II), with eligible par. being randomized to receive placebo or eltrombopag in each phase.
Pre-assignment Details: A total of 108 par. were randomized, of which 101 par. received at least 1 dose of study drug. A maximum of 6 cycles (with some exceptions) of chemotherapy with eltrombopag/placebo were allowed in each phase (either 21-day or 28-day cycle) followed by the 30 day Follow-up visit.
Groups:
- Phase I: 21-Day Cycle Placebo: Participants receiving gemcitabine on Day 1 and Day 8 plus carboplatin (G+Cb) or cisplatin (G+Cis) on Day 1 (Cis may be divided on Day 1 and Day 8) as a part of the 21-day chemotherapy cycle were administered placebo once daily for 5 days before and 5 days after Day 1 of Cycle 2 and subsequent chemotherapy cycles.
- Phase I: 21-Day Cycle Eltrombopag 100 mg: Participants receiving gemcitabine on Day 1 and Day 8 plus carboplatin (G+Cb) or cisplatin (G+Cis) on Day 1 (Cis may be divided on Day 1 and Day 8) as a part of the 21-day chemotherapy cycle were administered eltrombopag 100 milligrams (mg) once daily for 5 days before and 5 days after Day 1 of Cycle 2 and subsequent chemotherapy cycles.
- Phase I: 28-Day Cycle Placebo: Participants receiving gemcitabine on Day 1, Day 8 and Day 15 as a part of the 28-day chemotherapy cycle, were administered placebo once daily for 5 days before and 5 days after Day 1 of Cycle 2 and subsequent chemotherapy cycles.
- Phase I: 28-Day Cycle Eltrombopag 100 mg: Participants receiving gemcitabine on Day 1, Day 8 and Day 15 as a part of the 28-day chemotherapy cycle, were administered eltrombopag 100 mg once daily for 5 days before and 5 days after Day 1 of Cycle 2 and subsequent chemotherapy cycles.
- Phase II: Placebo: Participants receiving gemcitabine plus carboplatin or cisplatin as a part of 21-day chemotherapy cycle or gemcitabine alone as a part of the 28-day chemotherapy cycle, were administered placebo once daily for 5 days before and 5 days after Day 1 of each chemotherapy cycle (up to a maximum of 6 cycles).
- Phase II: Eltrombopag 100 mg: Participants receiving gemcitabine plus carboplatin or cisplatin as a part of 21-day chemotherapy cycle or gemcitabine alone as a part of the 28-day chemotherapy cycle were administered eltrombopag 100 mg once daily for 5 days before and 5 days after Day 1 of each chemotherapy cycle (up to a maximum of 6 cycles).
Period: Phase I (168 Days)
Arm/Group | Phase I: 21-Day Cycle Placebo | Phase I: 21-Day Cycle Eltrombopag 100 mg | Phase I: 28-Day Cycle Placebo | Phase I: 28-Day Cycle Eltrombopag 100 mg | Phase II: Placebo | Phase II: Eltrombopag 100 mg
Started | 3 | 9 | 4 | 10 | 0 | 0
Completed | 2 | 8 | 2 | 5 | 0 | 0
Not Completed | 1 | 1 | 2 | 5 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 0 | 0
Period: Phase II (168 Days)
Arm/Group | Phase I: 21-Day Cycle Placebo | Phase I: 21-Day Cycle Eltrombopag 100 mg | Phase I: 28-Day Cycle Placebo | Phase I: 28-Day Cycle Eltrombopag 100 mg | Phase II: Placebo | Phase II: Eltrombopag 100 mg
Started | 0 | 0 | 0 | 0 | 23 | 52
Ongoing | 0 | 0 | 0 | 0 | 1 | 0
Completed | 0 | 0 | 0 | 0 | 7 | 19
Not Completed | 0 | 0 | 0 | 0 | 16 | 33
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3 | 6
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 5 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 7 | 15
Not completed — Ongoing | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I: 28-Day Cycle Placebo: Participants receiving gemcitabine on Day 1, Day 8 and Day 15 as a part of 28-day chemotherapy cycle, were administered placebo once daily for 5 days before and 5 days after Day 1 of Cycle 2 and subsequent chemotherapy cycles.
- Phase I: 28-Day Cycle Eltrombopag 100 mg: Participants receiving gemcitabine on Day 1, Day 8 and Day 15 as a part of 28-day chemotherapy cycle, were administered eltrombopag 100 mg once daily for 5 days before and 5 days after Day 1 of Cycle 2 and subsequent chemotherapy cycles.
- Phase II: Placebo: Participants receiving gemcitabine plus carboplatin or cisplatin as a part of 21-day chemotherapy cycle or gemcitabine alone as a part of 28-day chemotherapy cycle, were administered placebo once daily for 5 days before and 5 days after Day 1 of each chemotherapy cycle (up to a maximum of 6 cycles).
- Phase II: Eltrombopag 100 mg: Participants receiving gemcitabine plus carboplatin or cisplatin as a part of 21-day chemotherapy cycle or gemcitabine alone as a part of 28-day chemotherapy cycle were administered eltrombopag 100 mg once daily for 5 days before and 5 days after Day 1 of each chemotherapy cycle (up to a maximum of 6 cycles).
- Total: Total of all reporting groups
Arm/Group | Phase I: 21-Day Cycle Placebo | Phase I: 21-Day Cycle Eltrombopag 100 mg | Phase I: 28-Day Cycle Placebo | Phase I: 28-Day Cycle Eltrombopag 100 mg | Phase II: Placebo | Phase II: Eltrombopag 100 mg | Total
Number analyzed (Participants) | 3 | 9 | 4 | 10 | 23 | 52 | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.3 (3.79) | 53.8 (11.27) | 61.8 (22.82) | 65.6 (8.41) | 64.4 (9.96) | 66.3 (8.98) | 64.1 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 3 | 3 | 13 | 23 | 50
  Male | 2 | 2 | 1 | 7 | 10 | 29 | 51
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 1 | 0 | 0 | 1 | 0 | 3
  White | 2 | 8 | 3 | 8 | 22 | 52 | 95
  Central/South Asian Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Japanese/East Asian Heritage/South East Asian | 0 | 0 | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE): Pre-therapy, On-therapy + 30 Days and Post-therapy in Phase I
Description: AEs are coded using the standard Medical Dictionary for Regulatory Activities (MedDRA) and were graded by the investigator according to National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE), version 4.0. AE is any untoward medical occurrence temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a MP. For marketed MPs, this also includes failure to produce expected benefits, abuse, or misuse. SAE event is any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or, is a congenital anomaly/birth defect.
Time Frame: From Cycle 1, Day 1 (C1D1) until at least 30 days post-investigational product discontinuation (longer for AEs considered related to study participation)
Population: Safety Population
Measure: Number; unit: Participants
Groups:
- 21-Day Cycle Placebo: Participants receiving gemcitabine on Day 1 and Day 8 plus carboplatin (G+Cb) or cisplatin (G+Cis) on Day 1 (Cis may be divided on Day 1 and Day 8) as a part of the 21-day chemotherapy cycle were administered placebo once daily for 5 days before and 5 days after Day 1 of Cycle 2 and subsequent chemotherapy cycles.
- 21-Day Cycle Eltrombopag 100 mg: Participants receiving gemcitabine on Day 1 and Day 8 plus carboplatin (G+Cb) or cisplatin (G+Cis) on Day 1 (Cis may be divided on Day 1 and Day 8) as a part of the 21-day chemotherapy cycle were administered eltrombopag 100 milligrams (mg) once daily for 5 days before and 5 days after Day 1 of Cycle 2 and subsequent chemotherapy cycles.
- 28-Day Cycle Placebo: Participants receiving gemcitabine on Day 1, Day 8 and Day 15 as a part of 28-day chemotherapy cycle, were administered placebo once daily for 5 days before and 5 days after Day 1 of Cycle 2 and subsequent chemotherapy cycles.
- 28-Day Cycle Eltrombopag 100 mg: Participants receiving gemcitabine on Day 1, Day 8 and Day 15 as a part of 28-day chemotherapy cycle, were administered eltrombopag 100 mg once daily for 5 days before and 5 days after Day 1 of Cycle 2 and subsequent chemotherapy cycles.
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Participants
  Any AE Pre-therapy | 3 | 8 | 4 | 9
  Any SAE Pre-therapy | 1 | 0 | 0 | 1
  Any AE On-therapy+30 days | 3 | 9 | 3 | 10
  Any SAE On-therapy+30 days | 1 | 5 | 1 | 2
  Any AE Post-therapy | 0 | 0 | 0 | 3
  Any SAE Post-therapy | 0 | 0 | 0 | 1
  Treatment-related AEs On-therapy+30 days | 2 | 3 | 1 | 6
  >=Grade 3 AEs On-therapy+30 days | 2 | 7 | 2 | 3
  Liver AEs On-therapy+30 days | 0 | 2 | 0 | 2
  Renal AEs On-therapy+30 days | 0 | 3 | 2 | 0
  Thromboembolic events On-therapy+30 days | 0 | 2 | 0 | 1
  Cardiac AEs On-therapy+30 days | 0 | 1 | 1 | 1
  Neutropenia On-therapy+30 days | 3 | 4 | 2 | 5
  Anemia On-therapy+30 days | 1 | 4 | 1 | 4
  Thrombocytopenia On-therapy+30 days | 2 | 3 | 3 | 3
  Leukopenia On-therapy+30 days | 1 | 2 | 2 | 3
  Thrombocytosis On-therapy+30 days | 2 | 2 | 1 | 2
  Platelet count increased On-therapy+30 days | 0 | 0 | 0 | 3

2. Primary Outcome: Number of Participants With Indicated Maximum Toxicity Grades for the Indicated Hematology Parameters, at Anytime Post-Baseline in Phase I
Description: Hematology parameters with a related NCI CTCAE (version 4.0) toxicity grading were summarized by toxicity grade at each scheduled assessment, the maximum toxicity grade reached by a participant post-Baseline was summarized. Hematology parameters included hemoglobin (increased), hemoglobin (anemia), lymphocytes (increased), lymphocytes (decreased), total absolute neutrophil count (ANC), platelets (PLT) and white blood cells (WBC). The Baseline value is defined as the value reported immediately prior to the administration of the first dose of chemotherapy in Cycle 1. Post-Baseline is defined as any time after the first dose of chemotherapy in Cycle 1 up to and including all follow-up visits. Only those participant available at the indicated time points were analyzed (represented by n=X,X,X,X in the category titles).
Time Frame: After Baseline (C1D1), on-treatment and 30 day follow-up
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Participants
  Hemoglobin (Increased), Grade 0, n=3,9,4,10 | 3 | 9 | 4 | 10
  Hemoglobin (Anemia), Grade 1, n=3,9,4,10 | 2 | 1 | 0 | 3
  Hemoglobin (Anemia), Grade 2, n=3,9,4,10 | 0 | 6 | 2 | 4
  Hemoglobin (Anemia), Grade 3, n=3,9,4,10 | 1 | 2 | 2 | 3
  Lymphocytes (Increased), Grade 0, n=3,9,4,10 | 3 | 8 | 4 | 10
  Lymphocytes (Increased), Grade 2, n=3,9,4,10 | 0 | 1 | 0 | 0
  Lymphocytes (Decreased), Grade 0, n=3,9,4,10 | 1 | 1 | 0 | 3
  Lymphocytes (Decreased), Grade 1, n=3,9,4,10 | 0 | 2 | 0 | 0
  Lymphocytes (Decreased), Grade 2, n=3,9,4,10 | 1 | 1 | 1 | 4
  Lymphocytes (Decreased), Grade 3, n=3,9,4,10 | 1 | 5 | 3 | 2
  Lymphocytes (Decreased), Grade 4, n=3,9,4,10 | 0 | 0 | 0 | 1
  Total ANC, Grade 0, n=1,2,1,2 | 0 | 2 | 1 | 0
  Total ANC, Grade 1, n=1,2,1,2 | 1 | 0 | 0 | 2
  PLT, Grade 0, n=3,9,4,10 | 0 | 1 | 0 | 2
  PLT, Grade 1, n=3,9,4,10 | 0 | 1 | 1 | 3
  PLT, Grade 2, n=3,9,4,10 | 0 | 3 | 1 | 3
  PLT, Grade 3, n=3,9,4,10 | 1 | 2 | 2 | 1
  PLT, Grade 4, n=3,9,4,10 | 2 | 2 | 0 | 1
  WBC, Grade 0, n=3,9,4,10 | 0 | 0 | 1 | 2
  WBC, Grade 1, n=3,9,4,10 | 0 | 1 | 0 | 2
  WBC, Grade 2, n=3,9,4,10 | 2 | 2 | 1 | 2
  WBC, Grade 3, n=3,9,4,10 | 1 | 5 | 2 | 3
  WBC, Grade 4, n=3,9,4,10 | 0 | 1 | 0 | 1

3. Primary Outcome: Number of Participants With Indicated Maximum Toxicity Grades for the Indicated Clinical Chemistry Laboratory Parameters, at Anytime Post-Baseline in Phase I
Description: Clinical chemistry laboratory parameters with a related NCI CTCAE (version 4.0) toxicity grading were summarized by toxicity grade at each scheduled assessment. Clinical chemistry laboratory parameters included albumin (Alb), urea/blood urea nitrogen (BUN), creatinine, aspartate amino transferase (AST), alanine amino transferase (ALT), alkaline phosphatase (ALP), total bilirubin (TB), direct bilirubin (DB) and international normalized ratio/Prothrombin time (PT). The Baseline value is defined as the value reported immediately prior to the administration of the first dose of chemotherapy in Cycle 1. Post-Baseline is defined as any time after the first dose of chemotherapy in Cycle 1 up to and including all follow-up visits. Only those participants available at the indicated time points were analyzed (represented by n=X,X,X,X in the category titles).
Time Frame: After Baseline (C1D1), on-treatment and 30 day follow-up
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Participants
  Alb, Grade 0, n=3,9,4,10 | 2 | 4 | 0 | 4
  Alb, Grade 1, n=3,9,4,10 | 1 | 2 | 2 | 5
  Alb, Grade 2, n=3,9,4,10 | 0 | 3 | 1 | 1
  Alb, Grade 3, n=3,9,4,10 | 0 | 0 | 1 | 0
  ALP, Grade 0, n=3,9,4,10 | 2 | 3 | 3 | 6
  ALP, Grade 1, n=3,9,4,10 | 1 | 5 | 1 | 1
  ALP, Grade 2, n=3,9,4,10 | 0 | 1 | 0 | 2
  ALP, Grade 3, n=3,9,4,10 | 0 | 0 | 0 | 1
  ALT, Grade 0, n=3,9,4,10 | 2 | 3 | 3 | 4
  ALT, Grade 1, n=3,9,4,10 | 1 | 4 | 1 | 5
  ALT, Grade 2, n=3,9,4,10 | 0 | 2 | 0 | 0
  ALT, Grade 3, n=3,9,4,10 | 0 | 0 | 0 | 1
  AST, Grade 0, n=3,9,4,10 | 2 | 4 | 2 | 5
  AST, Grade 1, n=3,9,4,10 | 1 | 3 | 2 | 3
  AST, Grade 2, n=3,9,4,10 | 0 | 1 | 0 | 1
  AST, Grade 3, n=3,9,4,10 | 0 | 1 | 0 | 1
  TB, Grade 0, n=3,9,4,10 | 3 | 5 | 3 | 8
  TB, Grade 1, n=3,9,4,10 | 0 | 2 | 0 | 0
  TB, Grade 2, n=3,9,4,10 | 0 | 2 | 1 | 0
  TB, Grade 3, n=3,9,4,10 | 0 | 0 | 0 | 2
  Ca (hypercalcemia), Grade 0, n=3,9,4,10 | 3 | 8 | 4 | 10
  Ca (hypercalcemia), Grade 1, n=3,9,4,10 | 0 | 1 | 0 | 0
  Ca (hypercalcemia), Grade 2, n=3,9,4,10 | 0 | 0 | 0 | 0
  Ca (hypercalcemia), Grade 3, n=3,9,4,10 | 0 | 0 | 0 | 0
  Ca (hypocalcemia), Grade 0, n=3,9,4,10 | 2 | 7 | 3 | 9
  Ca (hypocalcemia), Grade 1, n=3,9,4,10 | 1 | 1 | 0 | 0
  Ca (hypocalcemia), Grade 2, n=3,9,4,10 | 0 | 1 | 1 | 1
  Ca (hypocalcemia), Grade 3, n=3,9,4,10 | 0 | 0 | 0 | 0
  Creatinine, Grade 0, n=3,9,4,10 | 3 | 7 | 4 | 9
  Creatinine, Grade 1, n=3,9,4,10 | 0 | 1 | 0 | 1
  Creatinine, Grade 2, n=3,9,4,10 | 0 | 1 | 0 | 0
  Creatinine, Grade 3, n=3,9,4,10 | 0 | 0 | 0 | 0
  Glu (hyperglycemia), Grade 0, n=3,9,4,10 | 2 | 3 | 1 | 2
  Glu (hyperglycemia), Grade 1, n=3,9,4,10 | 0 | 4 | 2 | 4
  Glu (hyperglycemia), Grade 2, n=3,9,4,10 | 1 | 2 | 1 | 4
  Glu (hyperglycemia), Grade 3, n=3,9,4,10 | 0 | 0 | 0 | 0
  Glu (hypoglycemia), Grade 0, n=3,9,4,10 | 3 | 8 | 4 | 8
  Glu (hypoglycemia), Grade 1, n=3,9,4,10 | 0 | 0 | 0 | 1
  Glu (hypoglycemia), Grade 2, n=3,9,4,10 | 0 | 1 | 0 | 1
  Glu (hypoglycemia), Grade 3, n=3,9,4,10 | 0 | 0 | 0 | 0
  K (hyperkalemia), Grade 0, n=3,9,4,10 | 1 | 8 | 3 | 9
  K (hyperkalemia), Grade 1, n=3,9,4,10 | 2 | 1 | 0 | 0
  K (hyperkalemia), Grade 2, n=3,9,4,10 | 0 | 0 | 1 | 1
  K (hyperkalemia), Grade 3, n=3,9,4,10 | 0 | 0 | 0 | 0
  K (hypokalemia), Grade 0, n=3,9,4,10 | 2 | 5 | 3 | 7
  K (hypokalemia), Grade 1, n=3,9,4,10 | 1 | 3 | 1 | 3
  K (hypokalemia), Grade 2, n=3,9,4,10 | 0 | 0 | 0 | 0
  K (hypokalemia), Grade 3, n=3,9,4,10 | 0 | 1 | 0 | 0
  Na (hypernatremia), Grade 0, n=3,9,4,10 | 2 | 9 | 3 | 10
  Na (hypernatremia), Grade 1, n=3,9,4,10 | 1 | 0 | 1 | 0
  Na (hypernatremia), Grade 2, n=3,9,4,10 | 0 | 0 | 0 | 0
  Na (hypernatremia), Grade 3, n=3,9,4,10 | 0 | 0 | 0 | 0
  Na (hyponatremia), Grade 0, n=3,9,4,10 | 2 | 4 | 2 | 5
  Na (hyponatremia), Grade 1, n=3,9,4,10 | 1 | 4 | 0 | 5
  Na (hyponatremia), Grade 2, n=3,9,4,10 | 0 | 0 | 0 | 0
  Na (hyponatremia), Grade 3, n=3,9,4,10 | 0 | 1 | 2 | 0

4. Primary Outcome: Number of Participants With a Change From Baseline in Creatinine of >=26.5 Micromoles/Liter (UMOL/L) in Phase I
Description: The number of participants with at least 1 change from Baseline in creatinine, with an increase >=26.5 UMOL/L are reported. Creatinine clearance is estimated using the Cockcroft-Gault formula which is a method to approximate kidney function. The Baseline value is defined as the value reported immediately prior to the administration of the first dose of chemotherapy in Cycle 1.
Time Frame: After Baseline (C1D1), on-treatment and 30 day follow-up
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Participants | 0 | 3 | 1 | 2

5. Primary Outcome: Number of the Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status Scores at the Indicated Time Points in Phase I
Description: ECOG-Zubrod scores for the performance status are defined as follows: Score 0: Fully active, 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, 2: ambulatory and capable of all self-care but unable to carry out any work activities, 3: capable of only limited self-care, 4: completely disabled, 5: dead. The data is presented for the participants with the ECOG performance score at the indicated time points during the study.
Time Frame: Screening, C1D1, C2D1, C2D8, C2D15, C3D1, C4D1, C4D22, C5D1, C5D8, C6D1, C6D15
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Participants
  Screening, Score 0, n=3,9,4,10 | 3 | 5 | 1 | 3
  Screening, Score 1, n=3,9,4,10 | 0 | 3 | 3 | 7
  Screening, Score 2, n=3,9,4,10 | 0 | 1 | 0 | 0
  Screening, Score 3, n=3,9,4,10 | 0 | 0 | 0 | 0
  C1D1, Score 0, n=3,9,4,10 | 3 | 5 | 2 | 3
  C1D1, Score 1, n=3,9,4,10 | 0 | 3 | 2 | 7
  C1D1, Score 2, n=3,9,4,10 | 0 | 1 | 0 | 0
  C1D1, Score 3, n=3,9,4,10 | 0 | 0 | 0 | 0
  C2D1, Score 0, n=3,8,4,10 | 1 | 3 | 2 | 2
  C2D1, Score 1, n=3,8,4,10 | 1 | 4 | 1 | 8
  C2D1, Score 2, n=3,8,4,10 | 1 | 1 | 1 | 0
  C2D1, Score 3, n=3,8,4,10 | 0 | 0 | 0 | 0
  C2D8, Score 0, n=1,0,1,0 | 1 | NA — Zero participants were analyzed; therefore, a value was not available. | 0 | NA — Zero participants were analyzed; therefore, a value was not available.
  C2D8, Score 1, n=1,0,1,0 | 0 | NA — Zero participants were analyzed; therefore, a value was not available. | 0 | NA — Zero participants were analyzed; therefore, a value was not available.
  C2D8, Score 2, n=1,0,1,0 | 0 | NA — Zero participants were analyzed; therefore, a value was not available. | 1 | NA — Zero participants were analyzed; therefore, a value was not available.
  C2D8, Score 3, n=1,0,1,0 | 1 | NA — Zero participants were analyzed; therefore, a value was not available. | 0 | NA — Zero participants were analyzed; therefore, a value was not available.
  C2D15, Score 0, n=0,1,0,1 | NA — Zero participants were analyzed; therefore, a value was not available. | 0 | NA — Zero participants were analyzed; therefore, a value was not available. | 0
  C2D15, Score 1, n=0,1,0,1 | NA — Zero participants were analyzed; therefore, a value was not available. | 0 | NA — Zero participants were analyzed; therefore, a value was not available. | 1
  C2D15, Score 2, n=0,1,0,1 | NA — Zero participants were analyzed; therefore, a value was not available. | 1 | NA — Zero participants were analyzed; therefore, a value was not available. | 0
  C2D15, Score 3, n=0,1,0,1 | NA — Zero participants were analyzed; therefore, a value was not available. | 0 | NA — Zero participants were analyzed; therefore, a value was not available. | 0
  C3D1, Score 0, n=2,6,2,7 | 1 | 2 | 2 | 4
  C3D1, Score 1, n=2,6,2,7 | 1 | 2 | 0 | 3
  C3D1, Score 2, n=2,6,2,7 | 0 | 1 | 0 | 0
  C3D1, Score 3, n=2,6,2,7 | 0 | 1 | 0 | 0
  C4D1, Score 0, n=2,6,1,7 | 1 | 1 | 0 | 4
  C4D1, Score 1, n=2,6,1,7 | 1 | 3 | 1 | 3
  C4D1, Score 2, n=2,6,1,7 | 0 | 1 | 0 | 0
  C4D1, Score 3, n=2,6,1,7 | 0 | 1 | 0 | 0
  C4D22, Score 0, n=0,0,0,1 | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | 0
  C4D22, Score 1, n=0,0,0,1 | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | 0
  C4D22, Score 2, n=0,0,0,1 | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | 1
  C4D22, Score 3, n=0,0,0,1 | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | 0
  C5D1, Score 0, n=1,3,1,4 | 0 | 0 | 0 | 2
  C5D1, Score 1, n=1,3,1,4 | 1 | 1 | 1 | 2
  C5D1, Score 2, n=1,3,1,4 | 0 | 1 | 0 | 0
  C5D1, Score 3, n=1,3,1,4 | 0 | 1 | 0 | 0
  C5D8, Score 0, n=0,1,0,0 | NA — Zero participants were analyzed; therefore, a value was not available. | 0 | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available.
  C5D8, Score 1, n=0,1,0,0 | NA — Zero participants were analyzed; therefore, a value was not available. | 0 | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available.
  C5D8, Score 2, n=0,1,0,0 | NA — Zero participants were analyzed; therefore, a value was not available. | 0 | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available.
  C5D8, Score 3, n=0,1,0,0 | NA — Zero participants were analyzed; therefore, a value was not available. | 1 | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available.
  C6D1, Score 0, n=1,1,1,4 | 0 | 1 | 0 | 2
  C6D1, Score 1, n=1,1,1,4 | 1 | 0 | 1 | 2
  C6D1, Score 2, n=1,1,1,4 | 0 | 0 | 0 | 0
  C6D1, Score 3, n=1,1,1,4 | 0 | 0 | 0 | 0
  C6D15, Score 0, n=0,0,0,1 | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | 0
  C6D15, Score 1, n=0,0,0,1 | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | 1
  C6D15, Score 2, n=0,0,0,1 | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | 0
  C6D15, Score 3, n=0,0,0,1 | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | NA — Zero participants were analyzed; therefore, a value was not available. | 0

6. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Findings at Anytime Post-Baseline in Phase I
Description: A single safety 12-lead ECG was performed using a standard 12-lead ECG machine at screening and post-dose on C2D4. Three further ECGs were carried out at C2D8, C5D8 and C6D15. Change in ECG findings were categorized as 'Clinically significant change: favorable', 'No change or insignificant change' or 'Clinically significant change (CSC): unfavorable' as determined by the investigator. The Baseline value is defined as the value reported immediately prior to the administration of the first dose of chemotherapy in Cycle 1. Any time post-Baseline is defined by counting the participants under the worst result experienced post-Baseline. The best to worst order is 'Clinically significant change: favorable', 'No change or insignificant change', and then 'Clinically significant change (CSC): unfavorable. Only those participants available at the indicated time points were analyzed (represented by n=X,X,X,X in the category titles).
Time Frame: C2D4, C2D8, C5D8, C6D15
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Participants
  No change or insignificant change n=3,9,3,8 | 3 | 8 | 3 | 7
  CSC: unfavorable, n=3,9,3,8 | 0 | 1 | 0 | 1

7. Primary Outcome: Mean Day 1 Scheduled Pre-chemotherapy Platelet Count Evaluated Across Cycles 1 to 6 in Phase II
Description: Scheduled pre-chemotherapy platelet count is defined within each cycle as the platelet count assessment on which the decision to give or delay chemotherapy was made. This was averaged for each participant across Cycles 1 to 6 and a natural log transformation was applied to the average. The log-transformed values were compared between eltrombopag and placebo groups using an analysis of covariance (ANCOVA) model adjusting for cycle duration (21-day vs. 28-day), Baseline loge(platelet count) and part of study (part 1 or 2 of phase II). Only those participants available at indicated time points were analyzed (represented by n=X,X).
Time Frame: Day 1 (averaged across cycles 1 to 6)
Population: Intent-to Treat (ITT) Population: all randomized participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Giga (10^9) cells per liter (Gi/L)
Groups:
- Placebo: Participants receiving gemcitabine plus carboplatin or cisplatin as a part of 21-day chemotherapy cycle or gemcitabine alone as a part of 28-day chemotherapy cycle, were administered placebo once daily for 5 days before and 5 days after Day 1 of each chemotherapy cycle (up to a maximum of 6 cycles).
- Eltrombopag 100 mg: Participants receiving gemcitabine plus carboplatin or cisplatin as a part of 21-day chemotherapy cycle or gemcitabine alone as a part of 28-day chemotherapy cycle were administered eltrombopag 100 mg once daily for 5 days before and 5 days after Day 1 of each chemotherapy cycle (up to a maximum of 6 cycles).
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 48
Giga (10^9) cells per liter (Gi/L) | 193.34 (54.5) | 246.20 (49.8)
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag 100 mg; Test type: Superiority or Other; p = 0.103, ANCOVA; Percent difference = 21.1, 95% CI 2-sided [-3.9 to 52.5]

8. Secondary Outcome: Average Pre-chemotherapy Platelet Count at the Indicated Time Points in Phase I
Description: Pre-chemotherapy platelet count is defined for Cycle 1 as the platelet count (from central laboratory data) immediately preceding the first dose of chemotherapy within Cycle 1. For all subsequent cycles it is defined as the platelet count (from central laboratory data) immediately preceding, but limited to within 2 days prior to the first dose of chemotherapy at Day 1. For Group A, the chemotherapy cycle consisted of 21 days and for Group B, the chemotherapy cycle consisted of 28 days. Blood samples were collected to estimate platelet count at the following time points: Group A; Days 1 and 8 of Cycles 1 to 6. Group B; Days 1, 8 and 15 of Cycles 1 to 6. Only those participants available at indicated time points were analyzed (represented by n=X, X, X, X).
Time Frame: C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1,C4D8, C4D15, C5D1,C5D8, C5D15, C6D1,C6D8 and C6D15
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells per liter (G cells/L)
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Giga (10^9) cells per liter (G cells/L)
  C1 D1, n=3,9,4,9 | 239.3 (75.87) | 244.8 (48.47) | 223.8 (79.96) | 207.7 (65.51)
  C1 D8, n=3,6,3,9 | 180.7 (65.03) | 143.8 (33.88) | 144.0 (44.17) | 135.6 (52.52)
  C1 D15, n=0,0,2, 6 | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | 135.0 (84.85) | 97.5 (39.15)
  C2 D1, n=2,9,4,8 | 443.0 (168.29) | 545.8 (131.66) | 284.8 (84.11) | 473.3 (117.07)
  C2 D8, n=2,7,3,9 | 221.0 (94.75) | 335.6 (134.06) | 163.3 (35.30) | 333.0 (146.59)
  C2 D15, n=0,0,2,6 | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | 80.5 (0.71) | 142.7 (63.14)
  C3 D1, n=2,5,2,7 | 464.0 (36.77) | 484.6 (188.16) | 290.5 (180.31) | 435.4 (145.57)
  C3 D8, n=2,6,2,5 | 285.0 (39.60) | 292.2 (161.11) | 293.0 (199.40) | 465.2 (260.20)
  C3 D15, n=0,0,2,5 | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | 92.0 (45.25) | 183.4 (119.12)
  C4 D1, n=1,6,1,6 | 298.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 394.7 (154.28) | 609.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 388.3 (166.07)
  C4 D8, n=1,5,1,6 | 261.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 249.8 (122.29) | 335.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 366.5 (143.75)
  C4 D15, n=0,0,1,6 | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | 86.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 169.8 (120.56)
  C5 D1, n=1,2,1,4 | 245.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 529.5 (340.12) | 337.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 406.0 (174.89)
  C5 D8, n=1,1,1,4 | 144.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 123.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 311.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 403.5 (195.31)
  C5 D15, n=0,0,1,4 | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | 75.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 140.5 (42.93)
  C6 D1, n=1,1,1,3 | 512.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 123.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 440.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 360.3 (133.45)
  C6 D8, n=1,1,0,3 | 251.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 137.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | 428.0 (210.71)
  C6 D15, n=0,0,1,2 | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | NA (NA) — Zero participants were analyzed; therefore, a value was not available. | 113.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 101.0 (48.08)

9. Secondary Outcome: Average Within-subject Central Laboratory Platelet Count Prior to Scheduled Chemotherapy Across Cycles 2 to 6 in Phase I
Description: Within-subject platelet count for each participant was calculated by summing up the visit platelet counts from each of Cycles 1 to 6 and dividing it by the number of cycles in which the participant had data. The average within a treatment group was calculated by summing up the values from each participant within the treatment group and dividing it by the number of participants. These platelet counts are different from the pre-chemotherapy platelet counts for cycles where the chemotherapy dose was delayed. Average within-subject central laboratory platelet count prior to scheduled chemotherapy across Cycles 2 to 6 are summarized. Blood samples were collected on Days 1 and 8 of Cycles 2 to 6 for Group A and on Days 1, 8 and 15 from Cycles 2 to 6 for Group B to estimate the average within subject platelet count prior to scheduled chemotherapy. Only those participants available at the indicated time points were analyzed (represented by n=X,X,X,X in the category titles).
Time Frame: Day 1 (averaged across Cycles 2 to 6), Day 8 (averaged across Cycles 2 to 6)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells per liter (G cells/L)
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Giga (10^9) cells per liter (G cells/L)
  G+Cb, Day 1, n=1,3,0,0 | 296.80 (NA) — There was only one participant analyzed; therefore, SD could not be determined | 275.00 (144.253) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Day 8, n=1,3,0,0 | 235.00 (NA) — There was only one participant analyzed; therefore, SD could not be determined | 232.10 (77.329) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cis, Day 1, n=2,6,0,0 | 322.50 (82.731) | 526.00 (86.408) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cis, Day 8, n=2,6,0,0 | 326.85 (119.006) | 296.75 (119.342) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  Gm, Day1, n=0,0,4,9 | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 309.20 (123.133) | 442.79 (114.593)
  Gm, Day8, n=0,0,4,10 | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 204.20 (80.822) | 355.09 (148.539)
  Gm, Day15, n=0,0,3,10 | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 75.37 (18.292) | 164.24 (94.905)

10. Secondary Outcome: Platelet Count Nadir for Each Chemotherapy Cycle in Phase I
Description: Platelet nadir is defined as the lowest platelet count (from central laboratory data) reported after the first dose of chemotherapy within each cycle. Platelet count nadir is defined for each cycle. For Group A, the chemotherapy cycle consisted of 21 days and for Group B, the chemotherapy cycle consisted of 28 days. Blood samples were collected to estimate platelet nadir count at the following time points: Group A; Days 1, 4, 8, 15 and 17 of Cycles 1 and 2, at Days 1, 4, 8, 15 and 17 of Cycle 3 to 6. Group B; Days 1, 4, 8, 15, 22 and 24 of Cycles 1 to 6. Only those participants available at indicated time points were analyzed (represented by n=X, X, X, X).
Time Frame: Cycle 1 to Cycle 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells per liter (G cells/L)
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Giga (10^9) cells per liter (G cells/L)
  Cycle 1, n=3,9,4,10 | 30.67 (20.404) | 106.56 (113.338) | 60.50 (22.664) | 99.00 (75.700)
  Cycle 2, n=2,9,4,10 | 66.00 (9.899) | 122.44 (115.794) | 103.50 (62.952) | 135.50 (73.951)
  Cycle 3, n=2,7,2,7 | 47.00 (4.243) | 88.29 (71.807) | 78.50 (43.134) | 151.00 (111.946)
  Cycle 4, n=2,6,1,7 | 76.50 (4.950) | 87.50 (79.173) | 86.00 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 142.86 (91.908)
  Cycle 5, n=1,2,1,4 | 14.00 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 148.00 (182.434) | 75.00 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 113.25 (34.683)
  Cycle 6, n=1,1,1,4 | 24.00 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 13.00 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 110.00 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 122.75 (63.163)

11. Secondary Outcome: Central Laboratory Average Daily Area Under the Curve Platelet-time Course Across Cycles 2 to 6 in Phase I
Description: The average daily area under the platelet-time course was normalized by dividing the area under curve by total duration. This gives an estimated average platelet value over the time period from cycles 2 to 6. For 21-Day Cycle, the chemotherapy cycle consisted of 21 days and for 28-Day Cycle, the chemotherapy cycle consisted of 28 days. Blood samples were collected to estimate thrombocytes at the following time points: 21-Day Cycle; Days 1, 4, 8, 15 and 17 of Cycles 1 to 6. 28-Day Cycle; Days 1, 4, 8, 15, 22 and 24 of Cycles 1 to 6.
Time Frame: All assessments from Cycle 2 Day 1 to last assessment in Cycle 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells per liter (G cells/L)
Groups:
- 21-Day Cycle Eltrombopag 100 mg): Participants receiving gemcitabine on Day 1 and Day 8 plus carboplatin (G+Cb) or cisplatin (G+Cis) on Day 1 (Cis may be divided on Day 1 and Day 8) as a part of the 21-day chemotherapy cycle were administered eltrombopag 100 milligrams (mg) once daily for 5 days before and 5 days after Day 1 of Cycle 2 and subsequent chemotherapy cycles.
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg) | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Giga (10^9) cells per liter (G cells/L) | 260.97 (67.581) | 307.59 (95.110) | 183.68 (55.366) | 291.18 (99.718)

12. Secondary Outcome: Number of Participants With Thrombocytopenia of Grade 1, 2, 3 or 4 Across All the Chemotherapy Cycles in Phase I, Using Central Laboratory Platelet Count
Description: As per the CTCAE version 4.0, par. with a platelet count <LLN but >=75 x 10^9/L (Gi/L) were considered to have Grade 1 thrombocytopenia; par. with a platelet count <75Gi/L, but >=50Gi/L were considered to have Grade 2 thrombocytopenia; par. with a platelet count <50Gi/L, but >=25Gi/L were considered to have Grade 3 thrombocytopenia and par. with a platelet count <25Gi/L were considered to have Grade 4 thrombocytopenia. Blood samples were collected to estimate thrombocytes at the following time points: For Group A, the chemotherapy cycle consisted of 21 days and for Group B, the chemotherapy cycle consisted of 28 days. Blood samples were collected to estimate thrombocytes at the following time points: Group A; Days 1, 4, 8, 15 and 17 of Cycles 1 to 6. Group B; Days 1, 4, 8, 15, 22 and 24 of Cycles 1 to 6. Par. experiencing thrombocytopenia (Platelets <150Gi/L) at least once within a cycle are presented in the category title as n=X,X,X,X.
Time Frame: Cycle 1 to Cycle 6
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Participants
  Grade 1, n=3,9,4,10 | 0 | 2 | 1 | 3
  Grade 2, n=3,9,4,10 | 0 | 3 | 1 | 4
  Grade 3, n=3,9,4,10 | 1 | 1 | 1 | 0
  Grade 4, n=3,9,4,10 | 1 | 2 | 0 | 0
  Grade 0 / None, n=3,9,4,10 | 1 | 1 | 1 | 3

13. Secondary Outcome: Maximum Duration of Thrombocytopenia Across Cycles 2 to 6 in Phase I, Estimated Using Central Laboratory Platelet Counts
Description: Duration of thrombocytopenia is defined as a period of time in days from the first report of a platelet count with NCI CTCAE Grade 1-4 until the first subsequent report of a platelet count no longer meeting those criteria, regardless of rescue medication usage. It was assessed between Day 1 of Cycle 2 and up to and including any Conclusion/Early Withdrawal visit assigned to the same cycle for participants completing up to 6 cycles, and between Day 1 of Cycle 2 and up to and including the end of Cycle 6 for participants continuing beyond 6 cycles. The chemotherapy cycle for Group A was 21 days and for Group B was 28 days. Blood samples were collected to estimate thrombocytes at the following time points: Group A; Days 1, 4, 8, 15 and 17 of Cycles 2 to 6. Group B; Days 1, 4, 8, 15, 22 and 24 of Cycles 2 to 6.
Time Frame: Cycle 2 to Cycle 6
Population: Safety Population. Participants experiencing thrombocytopenia with subsequent increase in platelet count to >=150Gi/L are included.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 2 | 8 | 3 | 7
Days | 11.0 (4.24) | 10.6 (5.63) | 14.7 (7.77) | 13.4 (5.06)

14. Secondary Outcome: Central Laboratory Platelet Count for Time Taken to Reach Platelet Nadir for Each Chemotherapy Cycle in Phase I
Description: Platelet nadir is defined within each cycle as the lowest platelet count reported after the Day 1 chemotherapy dose. The time taken to reach platelet nadir is defined within each cycle. For Group A, the chemotherapy cycle consisted of 21 days and for Group B, the chemotherapy cycle consisted of 28 days. Blood samples were collected to estimate platelet nadir count at the following time points: Group A; Days 1, 4, 8, 15 and 17 of Cycles 1 to 6. Group B; Days 1, 4, 8, 15, 22 and 24 of Cycles 1 to 6. Only those participants available at indicated time points were analyzed (represented by n=X, X, X, X).
Time Frame: Cycle 1 to Cycle 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Days
  Cycle 1, n=3,9,4,10 | 15.7 (0.58) | 11.4 (5.53) | 13.8 (6.13) | 13.8 (4.73)
  Cycle 2, n=2,9,4,10 | 15.0 (1.41) | 12.9 (4.68) | 14.0 (5.72) | 19.2 (4.42)
  Cycle 3, n=2,7,2,7 | 15.0 (1.41) | 12.9 (3.02) | 23.5 (0.71) | 17.6 (4.50)
  Cycle 4, n=2,6,1,7 | 14.0 (0.00) | 13.5 (3.33) | 14.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined | 17.4 (6.16)
  Cycle 5, n=1,2,1,4 | 15.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined | 11.5 (6.36) | 14.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined | 21.5 (1.00)
  Cycle 6, n=1,1,1,4 | 16.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined | 14.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined | 23.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined | 15.5 (5.20)

15. Secondary Outcome: Time to Recovery From Platelet Nadir for Each Chemotherapy Cycle in Phase I, Estimated Using Central Laboratory Platelet Counts
Description: Platelet nadir is defined within each cycle as the lowest platelet count reported after the Day 1 chemotherapy dose. Time to recovery (TR) (>100Gi/L or >150Gi/L) from platelet nadir is defined within each cycle as the time in days from the platelet nadir to the time at which platelet count returns to >=100Gi/L or >=150Gi/L within the same cycle or up to and including Day 1 of the next cycle. For the last cycle in the study, time to recovery was calculated in the same manner but up to and including any Conclusion/Early Withdrawal visit which has been assigned to the same cycle. For Group A, the chemotherapy cycle consisted of 21 days and for Group B, the chemotherapy cycle consisted of 28 days. Blood samples were collected to estimate platelet count at: Group A; Days 1, 4, 8, 15 and 17 of Cycles 1 to 6. Group B; Days 1, 4, 8, 15, 22, and 24 of Cycles 1 to 6. Only those participants available at indicated time points were analyzed (represented by n=X, X, X, X).
Time Frame: Cycle 1 to Cycle 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Days
  TR(<100Gi/L to >=100Gi/L), Cycle 1, n=3,6,4,7 | 5.3 (0.58) | 7.2 (2.56) | 7.0 (0.00) | 7.7 (2.87)
  TR(<100Gi/L to >=100Gi/L), Cycle 2, n=2,5,3,4 | 6.5 (2.12) | 6.6 (3.65) | 6.0 (4.00) | 7.0 (5.10)
  TR(<100Gi/L to >=100Gi/L), Cycle 3, n=1,4,0,2 | 7.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 8.5 (3.70) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 6.0 (1.41)
  TR(<100Gi/L to >=100Gi/L), Cycle 4, n=1,4,1,2 | 2.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 6.5 (5.20) | 14.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 5.0 (2.83)
  TR(<100Gi/L to >=100Gi/L), Cycle 5, n=1,1,1,1 | 5.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 5.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 9.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 7.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined.
  TR(<100Gi/L to >=100Gi/L), Cycle 6, n=0,1,0,0 | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 7.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  TR(<150Gi/L to >=150Gi/L), Cycle 1, n=3,7,4,8 | 5.3 (0.58) | 7.6 (2.57) | 7.0 (0.00) | 8.5 (3.46)
  TR(<150Gi/L to >=150Gi/L), Cycle 2, n=2,4,3,5 | 6.5 (2.12) | 7.8 (2.99) | 9.0 (4.36) | 9.4 (4.28)
  TR(<150Gi/L to >=150Gi/L), Cycle 3, n=1,6,1,5 | 7.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 8.0 (2.97) | 7.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 6.2 (1.10)
  TR(<150Gi/L to >=150Gi/L), Cycle 4, n=1,4,1,4 | 8.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 7.8 (4.27) | 14.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 8.3 (3.95)
  TR(<150Gi/L to >=150Gi/L), Cycle 5, n=1,0,1,3 | 5.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 14.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 4.7 (2.52)
  TR(<150Gi/L to >=150Gi/L), Cycle 6, n=0,0,1,0 | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 5.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.

16. Secondary Outcome: Dose Intensity of Gemcitabine Plus Cisplatin (G+Cis)/Gemcitabine Plus Carboplatin (G+Cb) and Gemcitabine Across Chemotherapy Cycles 1 to 6 in Phase I
Description: Dose intensity of chemotherapy is defined as the actual dose of chemotherapy given as a percentage of the scheduled C1D1/C1D8 dose, as applicable, within this study: Cycle Dose Intensity (%) = Total Actual dose (mg/m^2) within Cycle *100/ Total Scheduled dose (mg/m^2) in Cycle 1; wherein Actual Dose (mg/m^2) = Actual dose (mg)/Body Surface Area reported on electronic case report form (eCRF).
Time Frame: Cycle 1 to Cycle 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Dose Intensity (%)
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 3 | 9 | 4 | 10
Dose Intensity (%)
  G+Cis, Gemcitabine, Cycle 1, n=2,5,0,0 | 100.0 (0.00) | 99.8 (0.45) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cis, Gemcitabine, Cycle 2, n=1,5,0,0 | 100.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 92.8 (24.83) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cis, Gemcitabine, Cycle 3, n=1,4,0,0 | 100.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 104.3 (8.50) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cis, Gemcitabine, Cycle 4, n=1,3,0,0 | 100.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 83.3 (28.87) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cis, Cisplatin, Cycle 1, n=2,6,0,0 | 100.0 (0.00) | 100.3 (1.03) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cis, Cisplatin, Cycle 2, n=1,6,0,0 | 100.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 102.8 (6.05) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cis, Cisplatin, Cycle 3, n=1,5,0,0 | 100.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 93.8 (24.34) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cis, Cisplatin, Cycle 4, n=1,4,0,0 | 100.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 100.3 (0.96) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cis, Cisplatin, Cycle 5, n=0,1,0,0 | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 50 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Gemcitabine, Cycle 1, n=1,2,0,0 | 99.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 100.0 (0.00) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Gemcitabine, Cycle 2, n=1,2,0,0 | 99.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 88.5 (17.68) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Gemcitabine, Cycle 3, n=1,2,0,0 | 99.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 100.0 (0.00) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Gemcitabine, Cycle 4, n=1,2,0,0 | 49.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 99.5 (0.71) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Gemcitabine, Cycle 5, n=1,1,0,0 | 99.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 74.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Gemcitabine, Cycle 6, n=1,1,0,0 | 99.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 74.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Carboplatin, Cycle 1, n=1,3,0,0 | 101.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 88.7 (14.05) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Carboplatin, Cycle 2, n=1,3,0,0 | 100.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 103.0 (5.20) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Carboplatin, Cycle 3, n=1,2,0,0 | 93.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 105.0 (5.66) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Carboplatin, Cycle 4, n=1,2,0,0 | 91.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 107.5 (2.12) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Carboplatin, Cycle 5, n=1,1,0,0 | 100.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 71.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  G+Cb, Carboplatin, Cycle 6, n=1,1,0,0 | 87.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 79.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  Gemcitabine, Cycle 1, n=0,0,1,7 | NA (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 100.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 94.7 (6.75)
  Gemcitabine, Cycle 2, n=0,0,1,7 | NA (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 100.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 85.0 (17.48)
  Gemcitabine, Cycle 3, n=0,0,1,4 | NA (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 100.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 79.5 (21.44)
  Gemcitabine, Cycle 4, n=0,0,0,4 | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 94.8 (4.11)
  Gemcitabine, Cycle 5, n=0,0,0,3 | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 93.7 (3.79)
  Gemcitabine, Cycle 6, n=0,0,0,3 | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | 72.7 (17.01)

17. Secondary Outcome: Number of Participants With at Least One Delay in Their Scheduled Dose of Chemotherapy in Any Cycle in Phase I
Description: Any delay in a scheduled dose of gemcitabine monotherapy or the combination of gemcitabine plus carboplatin or cisplatin was evaluated for eltrombopag and placebo treated participants.
Time Frame: All time on chemotherapy treatment
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | 21-Day Cycle Placebo | 21-Day Cycle Eltrombopag 100 mg | 28-Day Cycle Placebo | 28-Day Cycle Eltrombopag 100 mg
Number analyzed (Participants) | 1 | 3 | 4 | 10
Participants | 1 | 2 | 2 | 1

18. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE): Pre-therapy, On-therapy + 30 Days and Post-therapy in Phase II
Description: AE is any untoward medical occurrence temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a MP. For marketed MPs, this also includes failure to produce expected benefits, abuse, or misuse. SAE event is any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or, is a congenital anomaly/birth defect.
Time Frame: From first dose of investigational product (IP) until 30 days after discontinuation of IP (Longer for AEs related to study participation)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
Participants
  Any AE Pre Therapy | 0 | 1
  Any SAE Pre Therapy | 0 | 0
  Any AE On Therapy+30 days | 23 | 48
  Any SAE On Therapy+30 days | 12 | 16
  Any AE Post Therapy | 4 | 2
  Any SAE Post Therapy | 2 | 1
  Blood/lymphatic system disorders On-therapy+30 day | 21 | 40
  Thrombocytopenia On-therapy+30 days | 11 | 19
  Anemia On-therapy+30 days | 16 | 26
  Neutopenia On-therapy+30 days | 13 | 21
  Gastrointestinal disorders On-therapy+30 days | 12 | 25
  Blood Creatinine increased On-therapy+30 days | 3 | 2
  Vascular discorders On-therapy+30 days | 2 | 6
  Cardiac disorders On-therapy+30 days | 1 | 3
  Pulmonary embolism On-therapy+30 days | 0 | 1
  Portal vein thrombosis On-therapy+30 days | 1 | 0
  Deaths On-therapy+30 days | 9 | 13

19. Secondary Outcome: Number of Participants With Any Bleeding and Significant Bleeding as Assessed Using the World Health Organization (WHO) Bleeding Scale, Across Cycles 1-6 in Phase II
Description: The WHO Bleeding Scale is a measure of bleeding severity with the following grades: Grade 0=no bleeding; Grade 1=petechiae; Grade 2=mild blood loss; Grade 3=gross bleeding; Grade 4=debilitating blood loss. The WHO grades were further classified into the following categories: no bleeding=Grade 0; any bleeding=Grades 1 to 4; no clinically significant bleeding=Grades 0 to 1; clinically significant bleeding=Grades 2 to 4. Baseline is defined as the Day 1 assessment or the latest possible screening assessment. Across Cycles 1-6 included all assessments after first dose of chemotherapy up to the end of Cycle 6. Data exclused for participants taking drugs that affect platelet function or anticoagulants, from the time that the medication was started.
Time Frame: Screening, Day -5, Day 1 and 8 of Cycles 1 to 6 of 21-day cycle schedule, Day 1, 8 and 15 of cycles 1 to 6 of 28-day schedule, treatment withdrawal and 30-day follow-up
Population: ITT Population: Participants with at least one visit within the cycle.
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 12 | 35
Participants
  Grade 0 | 11 | 34
  Grade 1 | 1 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 1

20. Secondary Outcome: Number of Participants Requiring a Platelet Transfusion in Phase II
Description: Platelet transfusion was used as a rescue medication for the treatment of thrombocytopenia. Number of participants requiring a platelet transfusion during Cycles 1-6 was summarized and compared between treatment groups using a logistic regression model adjusted for cycle duration. Each cycle included assessments starting at Day 1 of the cycle.
Time Frame: Screening, Day -5, throughout cycles 1 to 6 and up to 30 days after IP discontinuation
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
Participants
  Cycle 1 | 0 | 4
  Cycle 2 | 2 | 3
  Cycle 3 | 0 | 2
  Cycle 4 | 1 | 1
  Cycle 5 | 0 | 0
  Cycle 6 | 0 | 0

21. Secondary Outcome: Number of Participants With at Least One Delay in Their Scheduled Dose of Chemotherapy in Any Cycle in Phase II
Description: Any delay in scheduled dose of gemcitabine monotherapy or the combination of gemcitabine plus carboplatin or cisplatin was evaluated for eltrombopag and placebo treated participants. Number of participants with any delay in dose during 21-day cycle or 28-day cycle, in part 1 or part 2 of the study is summarized and presented. Only those participants who actually received chemotherapy are included for the cisplatin and carboplatin components and all participants are included for the gemcitabine components (represented by n=X,X in the category titles).
Time Frame: Cycle 1 to Cycle 6
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
Participants
  Gemcitabine, 21-day cycle, n=11,22 | 5 | 7
  Carboplatin, 21-day cycle, n=4,12 | 4 | 5
  Cisplatin, 21-day cycle, n=7,9 | 1 | 2
  Gemcitabine, 28-day cycle, n=12,30 | 4 | 4

22. Secondary Outcome: Number of Participants With Any Dose Reduction in Their Scheduled Dose of Chemotherapy in Any Cycle in Phase II
Description: Dose reductions are required following potential drug-related toxicities. Number of participants with any dose reduction during 21-day cycle or 28-day cycle, in part 1 or part 2 of the study is summarized and presented. Only participants who actually received chemotherapy were included for the cisplatin and carboplatin components. All participants were included for the gemcitabine components.
Time Frame: Cycle 1 to Cycle 6
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
Participants
  Gemcitabine, 21-day cycle, n=11,22 | 7 | 6
  Carboplatin, 21-day cycle, n=4,12 | 2 | 2
  Cisplatin, 21-day cycle, n=7,9 | 0 | 3
  Gemcitabine, 28-day cycle, n=12,30 | 8 | 8

23. Secondary Outcome: Dose Intensity of Gemcitabine Plus Cisplatin(G+Cis)/Gemcitabine Plus Carboplatin (G+Cb) and Gemcitabine Across Chemotherapy Cycles 1-6 in Phase II
Description: Dose intensity of chemotherapy is defined as the actual dose of chemotherapy given as a percentage of the scheduled C1D1/C1D8 dose, as applicable, within this study: cycle Dose Intensity (%) = Total Actual dose (mg/m^2) within cycle *100/ Total Scheduled dose (mg/m^2) in Cycle 1; wherein Actual Dose (mg/m^2) = Actual dose (mg)/Body Surface Area reported on eCRF. The average chemotherapy dose intensity at Day 1 across Cycles 1 to 6, Day 8 across Cycles 1 to 6 and Day 15 across Cycles 1 to 6 was summarized and compared between treatment groups using an ANCOVA model adjusted for cycle duration and part of the study.
Time Frame: Cycle 1 to Cycle 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Dose Intensity (%)
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
Dose Intensity (%)
  Cycle 1, n=23,48 | 96.6 (10.65) | 97.9 (6.19)
  Cycle 2, n=19,37 | 113.1 (33.91) | 97.8 (24.99)
  Cycle 3, n=13,26 | 102.6 (42.20) | 98.7 (35.77)
  Cycle 4, n=11,19 | 96.6 (27.65) | 90.7 (30.00)
  Cycle 5, n=6,12 | 102.2 (31.88) | 81.3 (25.39)
  Cycle 6, n=5,7 | 84.4 (21.92) | 65.2 (25.48)
  Cycle 1-6, n=23,49 | 98.5 (18.26) | 94.6 (15.71)

24. Secondary Outcome: Number of Participants With Indicated Maximum Toxicity Grades for the Indicated Hematology Parameters, at Anytime Post-Baseline in Phase II
Description: Hematology parameters with a related NCI CTCAE (version 4.0) toxicity grading were summarized by toxicity grade at each scheduled assessment, the maximum toxicity grade reached by a participant post-Baseline was summarized. Hematology parameters included Hemoglobin (Hb) increased, Anemia, Lymphocyte count (Lym), platelet count, White Blood Cell count (WBC) and Total Absolute Neutrophil Count (Total ANC). The Baseline value is defined as the value reported immediately prior to the administration of the first dose of chemotherapy in Cycle 1. Post-Baseline is defined as any time after the first dose of chemotherapy in Cycle 1 up to and including all follow-up visits. participants with missing Baseline value were assumed to have normal Baseline value. Only those Participant available at the indicated time points were analyzed (represented by n=X,X in the category titles).
Time Frame: After baseline (C1D1), on-treatment and 30 day follow-up
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
Participants
  Hb (Increased), Grade 0, n=23,52 | 23 | 52
  Hb (Increased), Grade 1, n=23,52 | 0 | 0
  Hb (Increased), Grade 2, n=23,52 | 0 | 0
  Hb (Increased), Grade 3, n=23,52 | 0 | 0
  Hb (Increased), Grade 4, n=23,52 | 0 | 0
  Hb (Anemia), Grade 0, n=23,52 | 0 | 4
  Hb (Anemia), Grade 1, n=23,52 | 4 | 16
  Hb (Anemia), Grade 2, n=23,52 | 13 | 16
  Hb (Anemia), Grade 3, n=23,52 | 6 | 16
  Hb (Anemia), Grade 4, n=23,52 | 0 | 0
  Lym (Increased), Grade 0, n=23,52 | 22 | 47
  Lym (Increased), Grade 1, n=23,52 | 0 | 0
  Lym (Increased), Grade 2, n=23,52 | 1 | 2
  Lym (Increased), Grade 3, n=23,52 | 0 | 1
  Lym (Increased), Grade 4, n=23,52 | 0 | 0
  Lym (Decreased), Grade 0, n=23,52 | 1 | 7
  Lym (Decreased), Grade 1, n=23,52 | 3 | 10
  Lym (Decreased), Grade 2, n=23,52 | 8 | 14
  Lym (Decreased), Grade 3, n=23,52 | 9 | 16
  Lym (Decreased), Grade 4, n=23,52 | 2 | 3
  Total ANC, Grade 0, n=23,52 | 4 | 16
  Total ANC, Grade 1, n=23,52 | 1 | 4
  Total ANC, Grade2, n=23,52 | 3 | 17
  Total ANC, Grade 3, n=23,52 | 10 | 10
  Total ANC, Grade 4, n=23,52 | 5 | 3
  Platelet count, Grade 0, n=23,52 | 0 | 7
  Platelet count, Grade 1, n=23,52 | 4 | 9
  Platelet count, Grade 2, n=23,52 | 3 | 9
  Platelet count, Grade 3, n=23,52 | 6 | 15
  Platelet count, Grade 4, n=23,52 | 10 | 12
  WBC count, Grade 0, n=23,52 | 4 | 14
  WBC count, Grade 1, n=23,52 | 3 | 10
  WBC count, Grade 2, n=23,52 | 8 | 17
  WBC count, Grade 3, n=23,52 | 6 | 11
  WBC count, Grade 4, n=23,52 | 2 | 0

25. Secondary Outcome: Number of Participants With Indicated Worst-case Change From Baseline in Clinical Chemistry Laboratory Parameters Using CTCAE Toxicity Grading, at Anytime Post-Baseline in Phase II
Description: Clinical chemistry laboratory parameters with a related CTCAE (version 4.0) toxicity grading were summarized by toxicity grade at each scheduled assessment. Worst-case grade change of the laboratory parameters at anytime post-Baseline is presented as "Any grade increase", "Increase to Grade 3 or Grade 4". Clinical chemistry laboratory parameters included Albumin (Al), creatinine, AST, ALT, ALP, TB, Calcium hypercalcemia (CaHy)/hypocalcemia (CaHo), Glucose hyperglycemia (GluHy)/hypoglycemia (GluHo), Potassium hypernatremia (KHy)/hyponatremia (KHo) and Sodium hypernatremia (NaHy)/hyponatremia (NaHo). The Baseline value is defined as the value reported immediately prior to the administration of the first dose of chemotherapy in Cycle 1. Post-Baseline is defined as any time after the first dose of chemotherapy in Cycle 1 up to and including all follow-up visits. Only those Participant available at the indicated time points were analyzed (represented by n=X,X in the category titles).
Time Frame: After baseline (C1D1), on-treatment (collected on days 1 and 8 for subjects on 21-day cycle and on days 1, 8 and 15 for subjects on 28-day cycle) and 30 day follow-up
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
participants
  Al, Any grade increase, n=23,51 | 10 | 22
  Al, Increase to Grade 3, n=23,51 | 0 | 2
  Al, Increase to Grade 4, n=23,51 | 0 | 0
  ALP, Any grade increase, n=23,52 | 11 | 16
  ALP, Increase to Grade 3, n=23,52 | 1 | 2
  ALP, Increase to Grade 4, n=23,52 | 0 | 0
  ALT, Any grade increase, n=23,52 | 12 | 16
  ALT, Increase to Grade 3, n=23,52 | 3 | 2
  ALT, Increase to Grade 4, n=23,52 | 0 | 0
  AST, Any grade increase, n=23,52 | 11 | 15
  AST, Increase to Grade 3, n=23,52 | 3 | 2
  AST, Increase to Grade 4, n=23,52 | 0 | 0
  TB, Any grade increase, n=23,52 | 5 | 11
  TB, Increase to Grade 3, n=23,52 | 3 | 2
  TB, Increase to Grade 4, n=23,52 | 0 | 0
  CaHy, Any grade increase, n=23,51 | 0 | 1
  CaHy, Increase to Grade 3, n=23,51 | 0 | 0
  CaHy, Increase to Grade 4, n=23,51 | 0 | 0
  CaHo, Any grade increase, n=23,51 | 3 | 10
  CaHo, Increase to Grade 3, n=23,51 | 1 | 2
  CaHo, Increase to Grade 4, n=23,51 | 0 | 0
  Creatinine, Any grade increase, n=23,52 | 5 | 11
  Creatinine, Increase to Grade 3, n=23,52 | 1 | 0
  Creatinine, Increase to Grade 4, n=23,52 | 0 | 0
  GluHy, Any grade increase, n=23,52 | 13 | 31
  GluHy, Increase to Grade 3, n=23,52 | 2 | 3
  GluHy, Increase to Grade 4, n=23,52 | 0 | 0
  GluHo, Any grade increase, n=23,52 | 2 | 4
  GluHo, Increase to Grade 3, n=23,52 | 0 | 0
  GluHo, Increase to Grade 4, n=23,52 | 1 | 0
  NaHy, Any grade increase, n=23,52 | 0 | 2
  NaHy, Increase to Grade 3, n=23,52 | 0 | 0
  NaHy, Increase to Grade 4, n=23,52 | 0 | 0
  NaHo, Any grade increase, n=23,52 | 4 | 15
  NaHo, Increase to Grade 3, n=23,52 | 1 | 1
  NaHo, Increase to Grade 4, n=23,52 | 0 | 0
  KHy, Any grade increase, n=23,52 | 4 | 10
  KHy, Increase to Grade 3, n=23,52 | 1 | 1
  KHy, Increase to Grade 4, n=23,52 | 0 | 0
  KHo, Any grade increase, n=23,52 | 5 | 11
  KHo, Increase to Grade 3, n=23,52 | 1 | 4
  KHo, Increase to Grade 4, n=23,52 | 0 | 1

26. Secondary Outcome: Number of Participants With Change From Baseline in Creatinine of >=26.5 UMOL/L in Phase II
Description: Number of participants with at least 1 assessment of change from Baseline in creatinine, with increase >=26.5 UMOL/L are presented. The Baseline value is defined as the value reported immediately prior to the administration of the first dose of IP.
Time Frame: as for outcome 25
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
participants | 5 | 11

27. Secondary Outcome: Number of the Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status Scores at the Indicated Time Points in Phase II
Description: ECOG-Zubrod scores for the Performance Status were defined as follows: 0: Fully active, 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, 2: Ambulatory and capable of all self-care but unable to carry out any work activities, 3: Capable of only limited self-care, 4: Completely disabled, 5 and Unknown: Dead. The data is presented for the participants with the ECOG performance score at different time points during the study. Only those participants available at the indicated time points were analyzed (represented by n=X,X in the category titles).
Time Frame: Screening, C1D1, C2D1, C3D1, C4D1, C5D1, C6D1, C7D1, C8D1, C9D1, C10D1, C11D1, C12D1, C13D1, C14D1, C15D1, C16D1 and C17D1
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
participants
  Screening, Score 0, n=23,52 | 3 | 19
  Screening, Score 1, n=23,52 | 19 | 32
  Screening, Score 2, n=23,52 | 1 | 1
  C1D1, Score 0, n=23,49 | 4 | 20
  C1D1, Score 1, n=23,49 | 17 | 28
  C1D1, Score 2, n=23,49 | 0 | 1
  C1D1, Unknown, n=23,49 | 2 | 0
  C2D1, Score 0, n=19,36 | 4 | 16
  C2D1, Score 1, n=19,36 | 13 | 18
  C2D1, Score 2, n=19,36 | 2 | 2
  C3D1, Score 0, n=13,27 | 3 | 9
  C3D1, Score 1, n=13,27 | 9 | 16
  C3D1, Score 2, n=13,27 | 1 | 2
  C4D1, Score 0, n=11,19 | 4 | 8
  C4D1, Score 1, n=11,19 | 7 | 10
  C4D1, Score 2, n=11,19 | 0 | 1
  C5D1, Score 0, n=6,12 | 2 | 5
  C5D1, Score 1, n=6,12 | 4 | 6
  C5D1, Score 2, n=6,12 | 0 | 1
  C6D1, Score 0, n=6,7 | 2 | 3
  C6D1, Score 1, n=6,7 | 4 | 4
  C7D1, Score 0, n=3,2 | 1 | 0
  C7D1, Score 1, n=3,2 | 2 | 2
  C8D1, Score 0, n=2,1 | 1 | 0
  C8D1, Score 1, n=2,1 | 1 | 1
  C9D1, Score 1, n=2,1 | 2 | 1
  C10D1, Score1 n=2,0 | 2 | 0
  C11D1, Score 1, n=2,0 | 1 | 0
  C11D1, Score 2, n=2,0 | 1 | 0
  C12D1, Score 1, n=2,0 | 2 | 0
  C13D1, Score 0, n=2,0 | 1 | 0
  C13D1, Score 1, n=2,0 | 1 | 0
  C14D1, Score 0, n=2,0 | 1 | 0
  C14D1, Score 1, n=2,0 | 1 | 0
  C15D1, Score 1, n=2,0 | 2 | 0
  C16D1, Score 0, n=1,0 | 1 | 0
  C17D1, Score 2, n=1,0 | 1 | 0

28. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Findings at Cycle 1 Day 4 (2 to 6 Hours Post-dose) in Phase II
Description: A single safety 12-lead ECG was performed using a standard 12-lead ECG machine at screening and 2 to 6 hours post-dose on C1D4. Change in ECG findings were categorized as 'Clinically significant change (CSC): favorable', 'No change or insignificant change' or 'Clinically significant change (CSC): unfavorable' as determined by the investigator. The Baseline value is defined as the value reported immediately prior to the administration of the first dose of investigational product. Only those participants available at the indicated time points were analyzed (represented by n=X,X in the category titles).
Time Frame: C1D4
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
participants
  CSC favorable, n=22,45 | 0 | 2
  No change or insignificant change, n=22,45 | 20 | 42
  CSC: unfavorable, n=22,45 | 2 | 1

29. Secondary Outcome: Mean Day 8 Scheduled Pre-chemotherapy Platelet Counts Evaluated Across Cycles 1 to 6 in Phase II
Description: Scheduled pre-chemotherapy platelet count is defined within each cycle as the platelet count assessment on which the decision to give or delay chemotherapy was made. This was averaged for each subject across cycles 1 to 6 and a natural log transformation was applied to the average. The log-transformed values were compared between eltrombopag and placebo groups using an analysis of covariance (ANCOVA) model adjusting for cycle duration (21-day vs. 28-day), baseline loge(platelet count) and part of study (part 1 or 2 of phase II). The number of participants analyzed is the number with a Day 8 scheduled platelet count.
Time Frame: Day 8 (averaged across cycles 1 to 6)
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Giga (10^9) cells per liter (G cells/L)
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 20 | 42
Giga (10^9) cells per liter (G cells/L) | 162.18 (74.2) | 180.65 (59.1)
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag 100 mg; Test type: Superiority or Other; p = 0.407, ANCOVA; Percent difference = 12.9, 95% CI 2-sided [-15.6 to 51.1]

30. Secondary Outcome: Mean Day 15 Scheduled Pre-chemotherapy Platelet Counts Evaluated Across Cycles 1 to 6 in Phase II
Description: Scheduled pre-chemotherapy platelet count is defined within each cycle as the platelet count assessment on which the decision to give or delay chemotherapy was made. This was averaged for each subject across cycles 1 to 6 and a natural log transformation was applied to the average. The log-transformed values were compared between eltrombopag and placebo groups using an analysis of covariance (ANCOVA) model adjusting for cycle duration (21-day vs. 28-day), baseline loge(platelet count) and part of study (part 1 or 2 of phase II). The number of participants analyzed is the number with a Day 15 scheduled platelet count.
Time Frame: Day 15 (averaged across cycles 1 to 6)
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Giga (10^9) cells per liter (G cells/L)
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 9 | 22
Giga (10^9) cells per liter (G cells/L) | 95.10 (23.3) | 95.29 (52.1)
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag 100 mg; Test type: Superiority or Other; p = 0.802, ANCOVA; Percent difference = -4.4, 95% CI 2-sided [-33.5 to 37.4]

31. Secondary Outcome: Mean Within-subject Platelet Count Prior to Scheduled Chemotherapy Across Cycles 1 to 6 in Phase II
Description: Within-subject platelet count for each par. was calculated by summing up the visit platelet counts from each of Cycles 1 to 6 and dividing it by the number of cycles in which the par. had data. The average within a treatment group was calculated by summing up the values from each par. within the treatment 21-day cycle dividing it by the number of par. These platelet counts are different from the pre-chemotherapy platelet counts for cycles where the chemotherapy dose was delayed. Average within-subject central laboratory platelet count prior to scheduled chemotherapy across Cycles 1 to 6 are summarized. Blood samples were collected on Day 1 and 8 of Cycles 1 to 6 for 21-day cycle and on Day 1, 8 and 15 from Cycles 1 to 6 for 28-day cycle to estimate the average within subject platelet count prior to scheduled chemotherapy. Only those participants available at the indicated time points were analyzed (represented by n=X,X in the category titles).
Time Frame: Day 1, Day 8, Day 15 (all averaged across cycles 1 to 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells per liter (G cells/L)
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
Giga (10^9) cells per liter (G cells/L)
  Day1, n=23,48 | 221.0 (128.23) | 272.9 (120.92)
  Day 8, n=20,42 | 201.0 (143.75) | 207.4 (110.93)
  Day 15, n=9,22 | 97.5 (24.82) | 106.7 (54.73)

32. Secondary Outcome: Platelet Count Nadir for Each Chemotherapy Cycle in Phase II
Description: Platelet nadir is defined as the lowest platelet count reported after the first dose of chemotherapy within each cycle. Platelet count nadir is defined for each cycle. Blood samples were collected to estimate platelet nadir count at the following time points: 21-day cycle; Day 1, Day 4, Day 8, Day 15 and Day 17 of Cycles 1 to 6. 28-day cycle; Day 1, Day 4, Day 8, Day 15, Day 22, Day 24 of Cycles 1 to 6. Only those participants available at indicated time points were analyzed (represented by n=X, X).
Time Frame: Cycle 1 to Cycle 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells per liter (G cells/L)
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
Giga (10^9) cells per liter (G cells/L)
  Cycle 1, n=23,48 | 68.3 (47.74) | 77.2 (76.43)
  Cycle 2, n=19,37 | 61.5 (35.82) | 68.5 (48.92)
  Cycle 3, n=13,26 | 71.6 (53.80) | 84.7 (60.03)
  Cycle 4, n=11, 19 | 89.7 (116.73) | 86.9 (56.11)
  Cycle 5, n=6,11 | 51.7 (12.23) | 83.0 (58.63)
  Cycle 6, n=5,5 | 69.6 (62.76) | 136.6 (151.88)

33. Secondary Outcome: Average Daily Area Under the Platelet-time Course Across Cycles 1 to 6 in Phase II
Description: The average daily area under the platelet-time course was normalized by dividing the area under curve by total duration. This gives an estimated average platelet value over the time period from cycles 1 to 6. Blood samples were collected to estimate platelet count at the following time points: 21-day cycle; Days 1, 4, 8, 15 and 17 of Cycles 1 to 6. 28-day cycle; Days 1, 4, 8, 15, 22 and 24 of Cycles 1 to 6.
Time Frame: All assessments from Cycle 1 Day 1 to last assessment in Cycle 6
Population: ITT Population:Participants with platelet count data in at least one cycle in the study.
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells per liter (G cells/L)
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 48
Giga (10^9) cells per liter (G cells/L) | 153.00 (96.079) | 189.48 (79.583)

34. Secondary Outcome: Number of Participants With Thrombocytopenia of Grade 1, 2, 3 or 4 Across Cycles 1 to 6 in Phase II
Description: As per the CTCAE version 4.0, participants with a platelet count <LLN but >=75 x 10^9/L (Gi/L) were considered to have Grade 1 thrombocytopenia; participants with a platelet count <75Gi/L, but >=50Gi/L were considered to have Grade 2 thrombocytopenia; participants with a platelet count <50Gi/L, but >=25Gi/L were considered to have Grade 3 thrombocytopenia and participants with a platelet count <25Gi/L were considered to have Grade 4 thrombocytopenia. Blood samples were collected to estimate thrombocytes at the following time points: 21-day cycle; Days 1, 4, 8, 15 and 17 of Cycles 1 to 6. 28-day cycle; Days 1, 4, 8, 15, 22 and 24 of Cycles 1 to 6. Participants experiencing thrombocytopenia(Platelets <150Gi/L) at least once within cycle are presented in the category title as n=X,X.
Time Frame: Cycle 1 to Cycle 6
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 50
Participants
  Grade 1 | 4 | 9
  Grade 2 | 3 | 9
  Grade 3 | 8 | 15
  Grade 4 | 8 | 12
  None | 0 | 5

35. Secondary Outcome: Maximum Duration of Thrombocytopenia Across Cycles 1 to 6 in Phase II
Description: Duration of thrombocytopenia is defined as a period of time in days from the first report of a platelet count with NCI CTCAE Grade 1-4 until the first subsequent report of a platelet count no longer meeting those criteria, regardless of rescue medication usage. It was assessed between Day 1 of Cycle 2 and up to and including any Conclusion/Early Withdrawal visit assigned to the same cycle for participants completing up to 6 cycles, and between Day 1 of Cycle 2 and up to and including the end of Cycle 6 for participants continuing beyond 6 cycles. The chemotherapy cycle for 21-day cycle was 21 days and for 28-day cycle was 28 days. Blood samples were collected to estimate thrombocytes at the following time points: 21-day cycle; Days 1, 4, 8, 15 and 17 of Cycles 2 to 6. 28-day cycle; Days 1, 4, 8, 15, 22 and 24 of Cycles 2 to 6.
Time Frame: Cycle 1 to Cycle 6
Population: ITT Population: Participants with at least one period of thrombocytopenia where duration could be calculated.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 45
Days | 32.6 (20.31) | 23.5 (18.68)

36. Secondary Outcome: Time Taken to Reach Platelet Nadir for Each Chemotherapy Cycle in Phase II
Description: Platelet nadir is defined within each cycle as the lowest platelet count reported after the Day 1 chemotherapy dose. The time taken to reach platelet nadir is defined within each cycle. Blood samples were collected to estimate platelet nadir count at the following time points: 21-day cycle; Days 1, 4, 8, 15 and 17 of Cycles 1 to 6. 28-day cycle; Days 1, 4, 8, 15, 22 and 24 of Cycles 1 to 6. Only those participants available at indicated time points were analyzed (represented by n=X, X).
Time Frame: Cycle 1 to Cycle 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
Days
  Cycle 1, n=23,48 | 14.7 (4.85) | 15.7 (6.12)
  Cycle 2, n=19,37 | 15.1 (4.41) | 15.4 (3.62)
  Cycle 3, n=13,26 | 15.8 (5.64) | 14.3 (4.76)
  Cycle 4, n=11,19 | 15.4 (5.48) | 14.7 (5.19)
  Cycle 5, n=6,11 | 15.5 (6.38) | 13.8 (4.45)
  Cycle 6, n=5,5 | 13.6 (7.37) | 10.4 (6.31)
  Cycle 7,n=2,2 | 15.0 (0.00) | 7.5 (0.71)
  Cycle 8, n=2,1 | 12.5 (3.54) | 8.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined.
  Cycle 9, n=2,0 | 12.5 (3.54) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.

37. Secondary Outcome: Time to Recovery From Platelet Nadir for Each Chemotherapy Cycle in Phase II
Description: Platelet nadir is defined within each cycle as the lowest platelet count reported after the Day 1 chemotherapy dose. TR (>100Gi/L or >150Gi/L) from platelet nadir is defined within each cycle as the time in days from the platelet nadir to the time at which platelet count returns to >=100Gi/L or >=150Gi/L within the same cycle or up to and including Day 1 of the next cycle. For the last cycle in the study, time to recovery was calculated in the same manner but up to and including any Conclusion/Early Withdrawal visit which has been assigned to the same cycle. Blood samples were collected to estimate platelet count at: 21-day cycle; Days 1, 4, 8, 15 and 17 of Cycles 1 to 6. 28-day cycle; Days 1, 4, 8, 15, 22, and 24of Cycles 1 to 6. Time to recover censored if platelet count did not return to >=100/150 Gi/L. Censored results are excluded from calculation of summary statistics. Only those participants available at indicated time points were analyzed (represented by n=X, X).
Time Frame: Cycle 1 to Cycle 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Eltrombopag 100 mg
Number analyzed (Participants) | 23 | 52
Days
  TR(<100Gi/L to >=100Gi/L), Cycle 1, n=17, 32 | 8.1 (3.15) | 8.5 (3.70)
  TR(<150Gi/L to >=150Gi/L), Cycle 1, n=12, 29 | 9.3 (3.89) | 9.1 (3.26)
  TR(<100Gi/L to >=100Gi/L), Cycle 2, n=13, 24 | 9.9 (3.64) | 8.3 (2.56)
  TR(<150Gi/L to >=150Gi/L), Cycle 2, n=11, 21 | 10.5 (4.50) | 9.0 (3.31)
  TR(<100Gi/L to >=100Gi/L), Cycle 3, n=9, 12 | 10.1 (5.01) | 8.8 (3.16)
  TR(<150Gi/L to >=150Gi/L), Cycle 3, n=7, 14 | 10.4 (5.74) | 9.6 (3.43)
  TR(<100Gi/L to >=100Gi/L), Cycle 4, n=8, 10 | 10.0 (5.63) | 10.9 (4.77)
  TR(<150Gi/L to >=150Gi/L), Cycle 4, n=5, 11 | 10.2 (6.65) | 10.6 (5.39)
  TR(<100Gi/L to >=100Gi/L), Cycle 5, n=5,6 | 7.8 (1.10) | 8.8 (4.79)
  TR(<150Gi/L to >=150Gi/L), Cycle 5, n=2,4 | 8.0 (0.00) | 7.3 (1.50)
  TR(<100Gi/L to >=100Gi/L), Cycle 6, n=2,2 | 10.5 (6.36) | 8.5 (0.71)
  TR(<150Gi/L to >=150Gi/L), Cycle 6, n=2,1 | 10.5 (6.36) | 8.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined.
  TR(<100Gi/L to >=100Gi/L), Cycle 7, n=1,1 | 15.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 22.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined.
  TR(<150Gi/L to >=150Gi/L), Cycle 7, n=1,1 | 15.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | 22.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined.
  TR(<100Gi/L to >=100Gi/L), Cycle 8, n=1,1 | 14.0 (1.41) | 20.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined.
  TR(<150Gi/L to >=150Gi/L), Cycle 8, n=1,0 | 15.0 (NA) — There was only one participant analyzed; therefore, SD could not be determined. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  TR(<100Gi/L to >=100Gi/L), Cycle 9, n=2, | 14.0 (11.31) | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.
  TR(<150Gi/L to >=150Gi/L), Cycle 9, n=0, | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available. | NA (NA) — Zero participants were analyzed; therefore, mean and SD were not available.

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from Cycle 1, Day 1 for Phase I; and from the time the first dose of investigational product (IP) is administered for Phase II; up to 30 days following discontinuation of IP.
Groups:
- Phase I: 21-Day Cycle Eltrombopag: Participants receiving gemcitabine on Day 1 and Day 8 plus carboplatin (G+Cb) or cisplatin (G+Cis) on Day 1 (Cis may be divided on Day 1 and Day 8) as a part of the 21-day chemotherapy cycle were administered eltrombopag 100 milligrams (mg) once daily for 5 days before and 5 days after Day 1 of Cycle 2 and subsequent chemotherapy cycles.
- Phase II: Eltrombopag: Participants receiving gemcitabine plus carboplatin or cisplatin as a part of 21-day chemotherapy cycle or gemcitabine alone as a part of 28-day chemotherapy cycle were administered eltrombopag 100 mg once daily for 5 days before and 5 days after Day 1 of each chemotherapy cycle (up to a maximum of 6 cycles).
Arm/Group | Phase I: 21-Day Cycle Placebo | Phase I: 21-Day Cycle Eltrombopag | Phase I: 28-Day Cycle Placebo | Phase I: 28-Day Cycle Eltrombopag 100 mg | Phase II: Placebo | Phase II: Eltrombopag
Serious Adverse Events (participants affected / at risk) | 1/3 | 5/9 | 1/4 | 2/10 | 13/23 | 17/52
Other Adverse Events (participants affected / at risk) | 3/3 | 9/9 | 4/4 | 10/10 | 22/23 | 47/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: 21-Day Cycle Placebo (N=3) | Phase I: 21-Day Cycle Eltrombopag (N=9) | Phase I: 28-Day Cycle Placebo (N=4) | Phase I: 28-Day Cycle Eltrombopag 100 mg (N=10) | Phase II: Placebo (N=23) | Phase II: Eltrombopag (N=52)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 3
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Device damage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0
Seizure cluster (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: 21-Day Cycle Placebo (N=3) | Phase I: 21-Day Cycle Eltrombopag (N=9) | Phase I: 28-Day Cycle Placebo (N=4) | Phase I: 28-Day Cycle Eltrombopag 100 mg (N=10) | Phase II: Placebo (N=23) | Phase II: Eltrombopag (N=52)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 3 | 5 | 15 | 24
Leukopenia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 3 | 2 | 9
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 5 | 7
Neutropenia (Blood and lymphatic system disorders) | 3 | 5 | 2 | 6 | 13 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3 | 4 | 5 | 10 | 18
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 2 | 1 | 2 | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 4
Constipation (Gastrointestinal disorders) | 0 | 4 | 0 | 1 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 4 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 5
Nausea (Gastrointestinal disorders) | 1 | 6 | 1 | 1 | 2 | 10
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 3 | 5
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 4 | 8
Fatigue (General disorders) | 1 | 1 | 2 | 3 | 3 | 13
Oedema peripheral (General disorders) | 0 | 1 | 2 | 2 | 1 | 5
Pain (General disorders) | 0 | 0 | 0 | 1 | 2 | 2
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 5 | 3
Pyrexia (General disorders) | 1 | 1 | 2 | 0 | 4 | 3
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 5 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 2 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 2 | 3 | 4
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 6
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 3
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 5 | 6
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 3 | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 6 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 5
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1 | 2 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 4
Insomnia (Psychiatric disorders) | 0 | 2 | 2 | 0 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0
Hyperglycamia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 2
headache (Nervous system disorders) | 0 | 2 | 1 | 2 | 1 | 2
Platelet count increased (Investigations) | 0 | 0 | 0 | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.